CLINICAL TRIAL: NCT05796232
Title: Pharmacogenetics of Ketamine in Children Presenting Emesis and Recovery Agitation During Procedural Analgesia and Sedation Outside of the Operating Room
Brief Title: Pharmacogenetics of Ketamine in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 16/19
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Procedural Pain
Keywords: Procedural pain; Analgesia; Sedation; Children
MeSH Terms: conditions — Pain, Procedural; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The need to treat the children with painful diagnostic-therapeutic procedures has increased in the last years. There is evidence from a wide scientific literature that drugs available in the setting of procedural sedation and analgesia such as midazolam, fentanyl, nitrous oxide, ketamine and propofol are absolutely safe without a significant incidence of adverse effects, if administered by anaesthesiologists and also trained pediatricians outside the operating room. Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist that blocks glutamate excitatory effects. Ketamine's molecular mechanism is not restricted to the NMDA receptor. Several studies indicate interactions with a series of receptor systems, including opioid, cholinergic and dopaminergic receptors. Ketamine is a safe and effective drug during procedural analgesia and sedation applied to children outside the operating room. A recent multicenter study, showed that ketamine, without being associated with other analgesic or sedative drugs, is the drug regimen with the lowest risk of adverse effects during this procedures. Even though being safe, ketamine may cause some adverse effects. When ketamine is administered for procedural sedation outside the operating room, adverse effects more frequently recorded are emesis and recovery agitation, each with a prevalence of around 8%. Recovery agitation, defined as any abnormal behavioural response such as any combination of agitation, crying, hallucinations or nightmares after sedation, in some cases (around 1%) may be severe and leads to specific treatment, mainly benzodiazepines. Emesis and recovery agitation are minor adverse events, but both may be very unpleasant for the patient and may play a role in the perception of patients and their parents of the quality of sedation, especially in children who need repeated procedures. Identifying patients, particularly children with chronic illnesses and leukemia, at risk of emesis and recovery agitation may facilitate the choice of different drugs regimens, improving the quality of care. The aim of this study is the identification of genetic and epigenetic biomarkers useful to predict emesis and recovery agitation related to administration of ketamine for procedural sedation and analgesia applied to children and to correlate them with the pharmacokinetic profile.

ELIGIBILITY:
Inclusion Criteria:

1. Any child between 1 and 17 years of age needing sedation and analgesia for painful procedures, such as suture laceration, fracture reductions, burn medications, bone marrow aspiration, lumbar puncture, arthrocentesis, colonoscopy and others.
2. Use of intravenous ketamine as the sole sedative agent for the procedure.

Exclusion Criteria:

1. Children needing drugs other that ketamine for sedation, such as fentanyl, propofol, midazolam and dexmedetomidine .
2. Children with intellectual disability or with non typical neurodevelopment, such as children with autism.
3. Children with a history of allergy or hypersensibility to ketamine.
4. Parents limitations in language and understanding informed consent forms and procedures.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children between 1 and 17 years of age needing sedation and analgesia for painful procedures
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
To identify genetic variants associated with the development of emesis and recovery agitation after intravenous administration of ketamine | 10 minutes before procedural sedation
  Genotyping will be performed using Illumina Omni 2.5 + exome array. Biomarker identification will be performed considering the genetic contribution of variants focusing on 10 candidate genes relevant for the biotransformation (CYP2B6, CYP2C9, CYP3A4, CYP3A5, CYP2A6) and for pharmacodynamics (genes encoding for the NMDA receptor subunits: GRIN1 e GRIN2A-D) of ketamine, selected on the basis of literature. The independent variable associated with ketamine induced adverse effects will be the presence or not of functional variants in the candidate genes.

SECONDARY OUTCOMES:
To assess the maximum plasmatic concentration (Cmax) after intravenous administration of ketamine | 10 minutes before procedural sedation
  Ketamine and its main metabolite norketamine will be quantified in plasma through a method of liquid chromatography / tandem mass spectrometry. The pharmacokinetic parameters will be calculated using WinNonlin software.
To assess the area under the concentration curve from time 0 (AUC 0-last) after intravenous administration of ketamine | 10 minutes before procedural sedation
  Ketamine and its main metabolite norketamine will be quantified in plasma through a method of liquid chromatography / tandem mass spectrometry. The pharmacokinetic parameters will be calculated using WinNonlin software.
To assess the plasmatic half-life after intravenous administration of ketamine | 10 minutes before procedural sedation
  Ketamine and its main metabolite norketamine will be quantified in plasma through a method of liquid chromatography / tandem mass spectrometry. The pharmacokinetic parameters will be calculated using WinNonlin software.
To assess the plasmatic clearance defined as dose/AUC after intravenous administration of ketamine | 10 minutes before procedural sedation
  Ketamine and its main metabolite norketamine will be quantified in plasma through a method of liquid chromatography / tandem mass spectrometry. The pharmacokinetic parameters will be calculated using WinNonlin software.
To identify exosomal miRNAs linked to the development of emesis and recovery agitation after intravenous administration of ketamine | 10 minutes before procedural sedation
  Neuronal-derived exosomes will be isolated and miRNAs will be sequenced. miRNAs contained in neuronal-derived exosomes and associated with ketamine induced adverse effects will be quantified through next generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided